CLINICAL TRIAL: NCT02790099
Title: Double-blinded Randomized Controlled Study for Comparison of Surgical Rectus Sheath and Intrathecal Morphine for Postoperative Pain Control After Caesarean Section
Brief Title: Comparison of Surgical Rectus Sheath Block and Intrathecal Morphine
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Queen Mary Hospital, Hong Kong (Other)
Responsible Party: Principal Investigator, Lui Man Wa, Dr, Queen Mary Hospital, Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UW 14-345
Record Dates: First submitted 2016-05-21; First posted 2016-06-03 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Pain
Keywords: Pain; Postoperative pain control; Rectus sheath block; Intrathecal morphine; Caesarean section
MeSH Terms: conditions — Pain | interventions — Bupivacaine; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Rectus sheath block only (Experimental): Patient will be given surgical rectus sheath block postoperatively with 40ml of bupivacaine (2.5mg/mL) and 0.1ml of normal saline will be injected intrathecally at time of spinal anaesthesia.
  Interventions: Drug: Bupivacaine
- Intrathecal morphine group (Active Comparator): 0.1mg preservative free morphine will be injected intrathecally at time of spinal anesthesia and 40ml of normal saline will be injected as rectus sheath block.
  Interventions: Drug: Morphine
- Both intervention (Active Comparator): Patient will be given 0.1mg preservative free morphine intrathecally at time of spinal anaesthesia and surgical rectus sheath block with 40ml of bupivacaine (2.5mg/ml).
  Interventions: Drug: Bupivacaine; Drug: Morphine

INTERVENTIONS:
Drug: Bupivacaine — Surgical rectus sheath block will be performed by injection of 40ml bupivacaine (2.5mg/ml) before closure of rectus sheath during the operation.
  Other Names: Marcain
  Arms: Both intervention; Rectus sheath block only
Drug: Morphine — 0.1mg preservative free morphine will be injected intrathecally by anaesthesiologist at the time of spinal anaesthesia.
  Arms: Both intervention; Intrathecal morphine group

SUMMARY:
Pain is the main obstacle in delaying postoperative recovery and leads to prolonged hospital stay. Administration of intrathecal morphine during spinal anaesthesia can provide effective pain control. However, it is associated with significant side effects including nausea, vomiting and itchiness. Also, it is not suitable in all patients, for example, those with morphine allergy, or severe respiratory disease. Surgical rectus sheath block involves injection of local anaesthetic agents into the rectus sheath space before closure of the wound. It has been shown to provide adequate pain control with less systemic side effects. The aim of the study is to evaluate the effectiveness of surgical rectus sheath block and intrathecal morphine in post-Caesarean section pain control.

DETAILED DESCRIPTION:
The incidence of Caesarean section is increasing worldwide. Adequate post-operative analgesia is becoming an essential expectation of patients after Caesarean section. The process of recovery will be hindered by suboptimal pain control and eventually it will leads to immobilization and prolonged hospital stay.

Spinal anesthesia is usually the mode of anesthesia in pregnancy in view of increase general anesthetic risks. Intrathecal morphine can provide good pain control. However, pruritus can occur in up to 51% of patient, nausea and vomiting in up to 21%. Despite its significant side effects, there is an overall better patient satisfactory over use of intrathecal morphine. Due to its concern on respiratory depression, intrathecal morphine is not recommended in patients with severe respiratory disease, obstructive sleep apnoea or those receiving central nervous system depressants. As a result, there were numerous studies on alleviating the adverse effect and to search for other alternatives.

Rectus sheath block aims at blocking the terminal branches of 9th -12th intercostals nerve within the rectus sheath. They form rectus sheath plexus after piercing the posterior aspect of the rectus sheath and then branch into muscular and cutaneous branches. It can be given by anesthetist with or without ultrasound guidance. However, it involved additional time for administration of rectus sheath block and possibility of incorrect placement of catheter leading to ineffective analgesia.

On the contrary, surgical rectus sheath block was administrated by surgeon before closure of rectus sheath. It involves injection of local anesthetic in the rectus sheath space before closure of the wound under direct visual control. Surgical rectus sheath block was shown to be effective in postoperative pain control after transverse laparotomy in paediatrics patients. It was shown to be effective in postoperative pain control in Caesarean section without intrathecal morphine.

Surgical rectus sheath block may be a simple and safe alternative for intrathecal morphine. However, the evidence on its use in Obstetrics and Gynaecology was sparse and there is no study directly comparing the two different mode of analgesia. The aim of the study is to evaluate the use of surgical rectus sheath and intrathecal morphine for postoperative pain in Caesarean section; and its side effects profile.

ELIGIBILITY:
Inclusion Criteria:

* Planned for elective lower segment Caesarean section, using suprapubic transverse incision
* Willing and able to participate after the study has been explained
* Those understand either Cantonese, Putonghua or English

Exclusion Criteria:

* Patient with treatment for chronic pain
* History of narcotic abuse/ recreational drug use
* Allergy to opioids/ local anesthesia/ paracetamol/ tramadol/ non-steroidal anti-inflammatory drugs
* Patient with pre-eclampsia

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Actual)
Dates: Start 2014-09; Primary Completion 2016-01 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Pain score | at 12 hours postoperatively
  Pain score at rest and movement (elevation of head and shoulder at supine position), using visual analogue scale (0-10)

SECONDARY OUTCOMES:
Requirement of oral analgesics | within 24hours postoperatively
  Paracetamol 1gram four times a day on request basis will be prescribed. The number of time requiring paracetamol will be recorded. The need of additional analgesics will be recorded.
Time of mobilization | 3days postoperatively
  time of starting mobilization, defined as able to get out of bed without assistance
Side effect | 3days postoperatively
  side effects including itchiness, nausea/ vomiting, sedation
Pain score | Immediate postoperative
  Pain score at rest and movement (elevation of head and shoulder at supine position), using visual analogue scale (0-10), will be accessed at the recovery room after the operation.
Pain score | 4hours postoperatively
  Pain score at rest and movement (elevation of head and shoulder at supine position), using visual analogue scale (0-10)
Pain score | 8hrs postoperatively
  Pain score at rest and movement (elevation of head and shoulder at supine position), using visual analogue scale (0-10)
Pain score | 24hrs postoperatively
  Pain score at rest and movement (elevation of head and shoulder at supine position), using visual analogue scale (0-10)

CONTACTS AND LOCATIONS:
Overall Officials: Ernest H. Y. Ng, Study Chair — Queen Mary Hospital, Hong Kong
Locations (1):
- Department of Obstetrics and Gynaecology, Queen Mary Hospital, Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No
That's for patient privacy that individual participant data will not be available.

REFERENCES:
- [Background] Uchiyama A, Nakano S, Ueyama H, Nishimura M, Tashiro C. Low dose intrathecal morphine and pain relief following caesarean section. Int J Obstet Anesth. 1994 Apr;3(2):87-91. doi: 10.1016/0959-289x(94)90175-9. PMID 15636923
- [Background] Dahl JB, Jeppesen IS, Jorgensen H, Wetterslev J, Moiniche S. Intraoperative and postoperative analgesic efficacy and adverse effects of intrathecal opioids in patients undergoing cesarean section with spinal anesthesia: a qualitative and quantitative systematic review of randomized controlled trials. Anesthesiology. 1999 Dec;91(6):1919-27. doi: 10.1097/00000542-199912000-00045. No abstract available. PMID 10598635
- [Background] Sawi W, Choy YC. A comparative study of post operative analgesia, side effects profile and patient satisfaction using intrathecal fentanyl with and without morphine 0.1 mg in caesarean section. Middle East J Anaesthesiol. 2013 Feb;22(1):21-6. PMID 23833846
- [Background] Rozen WM, Tran TM, Ashton MW, Barrington MJ, Ivanusic JJ, Taylor GI. Refining the course of the thoracolumbar nerves: a new understanding of the innervation of the anterior abdominal wall. Clin Anat. 2008 May;21(4):325-33. doi: 10.1002/ca.20621. PMID 18428988
- [Result] Willschke H, Bosenberg A, Marhofer P, Johnston S, Kettner SC, Wanzel O, Kapral S. Ultrasonography-guided rectus sheath block in paediatric anaesthesia--a new approach to an old technique. Br J Anaesth. 2006 Aug;97(2):244-9. doi: 10.1093/bja/ael143. Epub 2006 Jun 23. PMID 16798774
- [Result] Niklasson B, Borjesson A, Carmnes UB, Segerdahl M, Ohman SG, Blanck A. Intraoperative injection of bupivacaine-adrenaline close to the fascia reduces morphine requirements after cesarean section: a randomized controlled trial. Acta Obstet Gynecol Scand. 2012 Dec;91(12):1433-9. doi: 10.1111/j.1600-0412.2012.01480.x. Epub 2012 Nov 1. PMID 22686512
- [Result] Crosbie EJ, Massiah NS, Achiampong JY, Dolling S, Slade RJ. The surgical rectus sheath block for post-operative analgesia: a modern approach to an established technique. Eur J Obstet Gynecol Reprod Biol. 2012 Feb;160(2):196-200. doi: 10.1016/j.ejogrb.2011.10.015. Epub 2011 Nov 21. PMID 22104479